CLINICAL TRIAL: NCT05156255
Title: Profile of Human Milk Oligosaccharides and FUT2 Polymorphism of Mothers in Indonesia: A Study on the Association Between Maternal Genotype-Phenotype Secretor Status and Short Chain Fatty Acid Profile Based on the Mother-Infant Genotype Pair
Brief Title: Profile of Human Milk Oligosaccharides and FUT2 Polymorphism of Mothers in Indonesia
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Klara Yuliarti, MD, Indonesia University
Other Study IDs: 21-08-0852
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Breastfeeding, Exclusive
Keywords: Human Milk Oligosaccharide; Short Chain Fatty Acid
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Breastmilk, whole blood, buccal cells, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Human milk oligosaccharides (HMOs), the third most abundant constituent of breastmilk, are known to have beneficial effects on infant immunity. Maternal genetic polymorphisms cause HMO variability. The FUT2 gene determines the secretor status, whereas the FUT3 gene is responsible for the expression of Lewis fucosyltransferase. Therefore, breastmilk can be classified to four groups according to the variation. To date, this variability has not been investigated in Indonesia. This study aims to evaluate the association between FUT2 gene polymorphism and 2'-Fucosyllactose (2'-FL) secretor phenotype. In addition, infant FUT2 gene polymorphism and short chain fatty acid (SCFA) profile from stool samples are also analysed.

DETAILED DESCRIPTION:
Eligible mother-infant pairs are explained about this study. Those willing to participate in this study are asked for written informed consent. Mothers are interviewed about their baseline characteristics, family pedigree, nutritional intake, and routine drug consumption. Infants are checked for their birth history. Both are measured for weight and height.

Four specimens are collected from the subjects:

1. Mother

   1. Breastmilk

      Breastmilk is expressed at 8-11 AM to avoid variability due to circadian rhythm. One breast is emptied, 30 mL of breastmilk is stored in a sterile container, and the rest is returned for feeding. Breastmilk is divided to five 2-mL cryovials and stored in a -80°C freezer. The remaining is stored in a -20°C freezer.
   2. Blood

   Blood samples (3 mL) are collected for DNA extraction.
2. Infant

   1. Buccal cells

      Buccal swab kits are used to obtain samples for DNA extraction.
   2. Stool

Stool specimens are collected at the age of four weeks in a sterile container and stored in a -80°C storage before short chain fatty acid profile analysis.

ELIGIBILITY:
Inclusion Criteria:

* Mother

  1. Minimum of 18 years old
  2. With term infants aged 2-5 weeks
  3. Exclusively breastfeed
  4. Healthy condition
  5. Agree to participate and sign the informed consent
* Infant

  1. Infant with mother who fulfil the eligibility criteria

Exclusion Criteria:

* Mother

  1. Has a Caucasian ancestor in two generations above
  2. Infant has multiple congenital anomalies
* Infant

  1. Has ever received antibiotics

Min Age: 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligible mothers and infants visiting the research site during recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Human milk oligosaccharides profile of Indonesian mothers | 1 day
  The concentration of 19 HMOs will be measured using high performance anion exhange chromatography with pulsed amperometric detection (HPAEC-PAD).
Proportion of FUT2 secretor genotype of mothers based on single nucleotide polymorphism (SNP) rs601338 | 1 day
  Sequencing of coding sequence (exon 2) of FUT2 gene will be performed using a previously known outer primer from the study by Lefebvre, et al (2020). The results will be aligned with database from www.ncbi.nlm.nih.gov to find the proportion of rs601338 among mothers.
Association between rs601338 FUT2 secretor genotype and 2'-FL secretor phenotype in mothers | 1 day
  The association between rs601338 FUT2 genotype (homozygous dominant, heterozygous, homozygous recessive) and 2'-FL concentration will be analysed using ANOVA test.

SECONDARY OUTCOMES:
Novel FUT2 polymorphism in Indonesian mothers | 1 day
  The sequencing result of exon 2 in the FUT2 gene will be aligned with database from www.ncbi.nlm.nih.gov to find novel variants. Additional information regarding existing variants will be browsed using the same database. The allele frequency of new variants will be calculated to determine new SNP.
Proportion of FUT2 secretor genotype of infants based on single nucleotide polymorphism (SNP) rs601338 | 1 day
  Sequencing of coding sequence (exon 2) of FUT2 gene will be performed using a previously known outer primer from the study by Lefebvre, et al (2020). The results will be aligned with database from www.ncbi.nlm.nih.gov to find the proportion of rs601338 among infants.
Novel FUT2 polymorphism in infant | 1 day
  The sequencing result of exon 2 FUT2 will be aligned with database from www.ncbi.nlm.nih.gov to find novel variants. Additional information regarding existing variants will be browsed using the same database. The allele frequency of new variants will be calculated to determine new SNP.
Profile of infant stool short chain fatty acid based on mother-infant FUT2 genotype pairs | 1 day
  The concentration of total short chain fatty acid, acetate, propionate, and butyrate in infant's stool will be measured using gas chromatography-mass spectrometry (GC-MS). Difference in the concentration between four mother-infant genotype pairs will be analysed using ANOVA test.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Yuliarti, MD, Principal Investigator — Dept of Pediatric, Faculty of Medicine, Universitas Indonesia/ Cipto Mangunkusumo General Hospital
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No